Athens, 23. 04. 2025

The effectiveness and efficacy of the combination of pharmacotherapy and cognitive

behavioral psychotherapy under the recovery perspective for patients with anxiety

disorders, depressive disorders, PTSD, obsessive-compulsive disorders, personality

disorders, bipolar disorders, schizophrenia and psychotic disorders.

Dr. phil., Dipl.-Psych., Stavroula Rakitzi

Clinical psychologist and cognitive behavioral psychotherapist

Private practice

ILISION 34 15771 Athens Greece

2111180571

6989766935

Stavroula@Rakitzi.onmicrosoft.com

Description linkedin Stavroula Rakitzi

ORCID: http://0000-0002-5231-6619

Polyxeni Georgila, M. D. Psychiatrist and cognitive behavioral psychotherapist

Private practice

ILISION 34 15771 Athens Greece

6932905259

polyxenigeorgila@gmail.com

Description linkedin Polyxeni Georgila

ORCID: http://0000-0003-3137-506X

Athens, 23/04/2025

1

## Informed consent to the research protocol

Dr. Stavroula Rakitzi, a clinical psychologist and cognitive behavioral psychotherapist, and Dr. Polyxeni Georgila, M.D., psychiatrist, will conduct a research protocol regarding the effectiveness and efficacy of the combination of pharmacotherapy with individual cognitive behavioral psychotherapy

The research protocol begins on 20. 05.2025. The tests will be administered before the therapy, after the therapy and in a follow-up after 6 months (24 weeks).

The test results will be used for statistical analysis to research the effectiveness and efficacy of the treatments. Results will be anonymous, and no personal data will be displayed from any individual participating in the groups. I will let you know about the results. My participation in these research protocol is voluntary. I certify that I have been informed of the above and that I agree with them.

| Name | Sig nature |
|------|------------|
| | Name |